CLINICAL TRIAL: NCT06425510
Title: Tech Enabled Functional Health: Bridging Primary Care Gaps for Older Latinos With Functional Disabilities in Underserved Communities
Brief Title: Using Technology to Improve Function for Older Latinos With Disabilities in Underserved Areas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2405230330
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Aging; Disability Physical
Keywords: self help devices; behavioral intervention; assistive technology; primary health care; community health workers; older Latinos

STUDY DESIGN:
Intervention Model Description: Social Cognitive Theory
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (VIVE-AT) - Translation: Living the Advantages of Technological Assistance (Experimental): The VIVE-AT program consists of a six-week, once-a-week, 2-hour group educational intervention guided by the social cognitive model. It is facilitated by primary care and community health workers in a primary healthcare clinic. The intervention aims to teach older Latinos self-management strategies to increase the adoption and use of assistive technology devices that enhance their function in daily activities. VIVE-AT is designed to support behavioral change by providing up to five assistive technology devices to participants, along with information, instruction, demonstration, action planning, and guided practice in using the devices.
  Interventions: Behavioral: Translation: Living the Advantages of Technological Assistance (VIVE-AT)
- Waitlist Control (Active Comparator): Participants in the waitlist control group will receive weekly attention calls providing general health advice during the 6-week intervention period. They will also receive usual care for the initial 6 months post-randomization, followed by crossover to the VIVE-AT intervention.
  Interventions: Other: Attention calls

INTERVENTIONS:
Behavioral: Translation: Living the Advantages of Technological Assistance (VIVE-AT) — It comprises 2-hour small group sessions of 8-10 participants, once a week, for six weeks of participatory discussions, experiential learning, multimodal instructions, and demonstration and practice with selected assistive technology devices (ATDs). The content of the VIVE-AT weekly sessions is as follows: Week 1 - Introduction to ATDs, funding, and resources; Week 2 - ATDs for self-care and toilet use; Week 3 - ATDs for mobility; Week 4 - ATDs for dressing; Week 6 - ATDs for cooking and home tasks. Each session is designed with the following components: monitoring of participants' weekly goals; providing information on ATDs, resources, and services; reflection on the advantages and disadvantages of using these ATDs; hands-on practice with selected ATDs; goal setting and addressing barriers to using ATDs. Group sessions will incorporate visual aids, including modeling and videos of older individuals using ATDs accessed through an AT web app in a tablet provided by this project.
  Arms: (VIVE-AT) - Translation: Living the Advantages of Technological Assistance
Other: Attention calls — Ten minutes of attention calls, once a week for six weeks, to the waitlist control participants will offer general health advice on topics like nutrition, exercise, sleep, stress, and social connections. These calls emphasize participant well-being without touching upon the specific VIVE-AT content, maintaining a clear distinction from the intervention group.
  Arms: Waitlist Control

SUMMARY:
This project aims to test a culturally appropriate assistive technology (AT) intervention called VIVE-AT to help older Latinos with disabilities improve their function and quality of life. The researchers will first refine the VIVE-AT program based on feedback from a Community Advisory Board and focus groups with older Latinos with disabilities. Then, 76 older Latinos with disabilities will be recruited from a primary care clinic serving low-income communities in Puerto Rico. They will be randomly assigned to either receive the VIVE-AT intervention in the primary care clinic or be placed on a waitlist with regular phone calls. All participants will continue to receive standard care at the clinic.

DETAILED DESCRIPTION:
Functional disabilities (FDs), defined as difficulties in performing daily activities, constitute a significant public health problem associated with increased dependency, poor health outcomes, diminished quality of life, institutionalization, and premature death. Older Latinos residing in Puerto Rico (PR) are disproportionately affected by FDs, with one of the highest rates of FDs (58%) in the US and its territories. Research has demonstrated positive outcomes from employing assistive technology (AT) devices, such as jar openers, sock aids, and canes, among older adults with FDs, thereby enhancing their functioning, participation, and capacity to remain at home or in the community for a longer period. However, Latinos are among the least likely to utilize AT. Given the dearth of culturally competent assistive technology interventions for Latinos, along with the scarcity of rehabilitation professionals and assistive technology services in primary healthcare facilities, this project leverages preliminary data from a prior study that assessed the feasibility of the Viviendo las Ventajas de la Asistencia Tecnológica; (VIVE-AT for short; Living the Advantages of Assistive Technologies) intervention. The specific aims of this project are to:

1. refine the protocol of the VIVE-AT to align with the unique needs of the primary health care clinic;
2. assess the efficacy of the VIVE-AT in comparison to a waitlist control arm, in decreasing FDs and improving the quality of life among Latinos aged ≥65 years post-intervention and at six months;
3. evaluate whether proposed mechanisms of change in FDs, specifically knowledge of AT, motivation for using AT, self-efficacy for using AT, and use of AT, account for the reduction in FDs post-intervention.

To achieve these aims, the interdisciplinary team of this project will first refine the intervention based on recommendations from participants in the feasibility study, as well as input from the Community Advisory Board and older Latinos with FDs through iterative focus groups (Aim 1). Subsequently, 76 older Latinos with physical FDs recruited from a primary health care facility serving low-income communities in PR will be randomly assigned to either the VIVE-AT intervention group (n=38) or a waitlist + attention calls controlled condition group (n=38) to assess its efficacy and mechanisms of change (Aims 2 and; 3). All participants will receive standard usual care at the primary health care center. Participants in the intervention group will attend a weekly, two-hour group session for 6 weeks, facilitated by trained healthcare workers, focusing on self-management of FDs through AT. Additionally, participants will receive up to five AT devices tailored to their specific functional disabilities needs, along with training on their usage. All participants will be assessed at baseline, post-intervention, and six months after intervention. The goals of the VIVE-AT are to encourage participants to use AT devices to self-manage their FDs and improve their quality of life. This approach will contribute to scientific knowledge and inform a subsequent scalable multisite Hybrid Type I Randomized Controlled Trial designed to evaluate its effectiveness in reducing physical function disabilities among older Latinos in primary healthcare settings in the U.S. and P.R.

ELIGIBILITY:
Inclusion Criteria:

* Spanish speaking Latino adults ≥65 years
* With a physical function impairment (PROMIS-HAQ T-Score ≤45)
* Living independently in the community (not requiring supervision to perform their daily living activities)
* Self-reported ability to participate in a 6 weeks of group intervention
* Having no plans to move for the next 12 months

Exclusion Criteria:

* Currently residing in a nursing or group home
* Receiving home healthcare services
* Having a significant cognitive impairment as evidenced by a score ≤23 in the Mini Mental State Examination (MMSE)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Physical Function as Assessed by the PROMIS Short Form v2.0 - Physical Function 24a (PROMIS-HAQ) | Baseline, at the end of the intervention (6 weeks), and at 6 months post-intervention
  This is a patient-reported outcome measure designed to assess physical FDs in adults across the categories of dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, errands, and chores. It comprises 20 items on a 5-point Likert-type scale, ranging from 5 "without difficulty" to 1 "unable to do".
Quality of Life as Assessed by PROMIS Scale v1.2 - Global Health | Baseline, at the end of the intervention (6 weeks), and at 6 months post-intervention
  This is a 10-item health-related quality of life measure with five domains: physical health, pain, fatigue, mental health, and social health, along with an overall health assessment. It also includes two subscales: Global Mental Health (GMH) and Global Physical Health (GPH).

SECONDARY OUTCOMES:
Use of Assistive Technology Devices as Assessed by Assistive Technology Awareness Scale (ATUAS) | Baseline, at the end of the intervention (6 weeks), and at 6 months post-intervention
  The ATUAS assesses participants' knowledge of 44 assistive technology devices. Participants are presented with photographs and names of the devices and asked if they possess each item. If the answer is 'No,' further questions will determine whether they use it (code 2) or not (code 1), are aware of its existence (code 3), or neither (code 4). Responses will be recoded into two categories: used (code 2) and not used (codes 1, 3, and 4) to calculate assistive technology device usage.
Assistive Technology Knowledge as Assessed by Assistive Technology Use and Awareness Scale (ATUAS) | Baseline, at the end of the intervention (6 weeks), and at 6 months post-intervention
  The ATUAS assesses participants' knowledge of 44 assistive technology devices. Participants are presented with photographs and names of the devices and asked if they possess each item. If the answer is 'No,' further questions will determine whether they use it (code 2) or not (code 1), are aware of its existence (code 3), or neither (code 4). Assistive technology knowledge is assessed by re-coding the answer for each assistive technology into two categories: aware (codes 1, 2, 3) versus not aware (code 4).
Motivation to Use Assistive Technology as Assessed by Attitudes Towards Assistive Device Scale (AADS) | Baseline, at the end of the intervention (6 weeks), and at 6 months post-intervention
  The AADS consists of 12 items designed to measure older adults' attitudes (motivation), including the substitution of care, the financial aspect of care, and the effect on privacy. It utilizes a Likert scale with 5 points, ranging from 5 (totally agree) to 1 (totally disagree), with interval scores ranging from 12 to 60. A high score indicates a positive attitude.
Intention to Use Assistive Technology as Assessed by Intention to Use Assistive Device Scale | Baseline, at the end of the intervention (6 weeks), and at 6 months post-intervention
  This measure consists of three items presenting increasing levels of intention (motivation) to use assistive technology devices. It employs a 5-point Likert scale, ranging from 1 (I do not have the intention to do this at all) to 5 (I certainly have the intention to do this). The total score ranges from 3 to 15; higher scores indicate a strong intention to use assistive technology devices.
Self-efficacy as Assessed by Self-efficacy Regarding Assistive Device Use | Baseline, at the end of the intervention (6 weeks), and at 6 months post-intervention
  This measure assesses self-efficacy for using assistive technology devices with three items, each representing increasing barriers. The interval scale ranges from 3 to 15; a higher score indicates higher self-efficacy.

OTHER OUTCOMES:
Participation rates | At the end of the intervention (6 weeks)
  The percent of eligible older Latinos who were enrolled (goal: ≥ 80%)
Retention rates | At the end of the intervention (6weeks) and at 6 months post-intervention
  The percent of older Latinos who complete the study measures at the end of the intervention and at 6 months post-intervention (goal: ≥ 80%).
Attrition rates | At the end of the intervention (6 weeks) and 6 months post-intervention
  The percent of participants who drop out or are lost to follow-up at the end of the intervention and at 6 months post-intervention, with reasons recorded when known (goal: ≤ 20%).
Completion rates | At 6 months post-intervention
  The percent of participants completing at least 4 of 6 group sessions (goal: ≥ 80%).
Acceptability as Assessed by Acceptability: Assessment will be conducted using the Intervention Acceptability and Implementation Questionnaire | At the end of the intervention (6 weeks)
  This questionnaire is based on the key dimensions outlined in the Theoretical Framework of Acceptability, which include affect, burden, perceived effectiveness, ethicality, coherence, opportunity costs, and self-efficacy. It features open-ended questions to further explore suggested improvements, identify successful components, and understand contextual issues that influenced the implementation of the intervention in primary care clinic, all based on the Practical Robust Implementation and Sustainability Model (PRISM). The goal is to achieve a mean satisfaction level of ≥ 80%.
Cost | Baseline, during the intervention, at the end of the intervention (6 weeks), and at 6 months post-intervention
  The researchers will document total intervention costs, costs per participant, and marginal costs related to changes in FDs PROMIS-HAQ T-scores, valuing resources at competitive market rates. Costs will be estimated in constant dollars using the Prospective Payment System Index. Key resource categories include participant recruitment, intervention preparation, labor costs, training, supervision, and materials. The researchers will distinguish between research-based and intervention costs. Emergency room visits, their costs, reasons, and institutional costs (hospitalizations) will be tracked. Primary care physician visits will be documented over 32 weeks (including a 6-week intervention and 6-month follow-up). Additionally, the researchers will analyze mortality incidence during the intervention and the subsequent 32 weeks. Data will be sourced from the primary care clinic for all participants, with detailed documentation of activities and resources used throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puerto Rico Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
De-identified quantitative data that can be publicly shared will be formatted for widely available statistical packages such as R, Statistical Package for the Social Sciences (SPSS), STATA, and Statistical Analysis System (SAS). All shared study materials, data, and metadata will be made publicly available through the University of Puerto Rico Institutional Repository at the University of Puerto Rico Institutional Digital Repository website at https://repositorio.upr.edu/. Data will be assigned a Digital Object Identifier (DOI) and searchable via the University of Puerto Rico Institutional Repository and other search engines.
Supporting Information: Study Protocol, SAP
Time Frame: Data and metadata will be deposited into the repository at the time of publication or by the end of the project period, whichever comes first. Data will be preserved for three years following the end of the grant period.
Access Criteria: The study's Individual Participant Data (IPD) would be accessible to the academic community and the public. This repository serves as a digital storage site for the scientific and creative work of the University of Puerto Rico. They will be able to access all shared study materials, data, and metadata. To access the repository, users can visit the University of Puerto Rico Digital Institutional Repository website at https://repositorio.upr.edu. The repository allows for the searching and browsing of content, which includes faculty research works.
URL: https://repositorio.upr.edu/